CLINICAL TRIAL: NCT05536323
Title: Comparison of the Incidence of Hypotension in Bolus Versus Continuous Administration of Remimazolam During Anesthesia Induction
Brief Title: Bolus Versus Continuous Remimazolam for Anesthetic Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Eunah Cho, MD, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RMZ_bolcon
Record Dates: First submitted 2022-09-05; First posted 2022-09-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Hypotension on Induction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus (Experimental): Anesthetic induction with bolus remimazolam administration
  Interventions: Drug: Remimazolam bolus
- Continuous (Experimental): Anesthetic induction with continuous remimazolam administration
  Interventions: Drug: Remimazolam continuous

INTERVENTIONS:
Drug: Remimazolam bolus — Remimazolam bolus 0.14-0.33 mg/kg 0.25-0.33 mg/kg, <40 years 0.19-0.25 mg/kg, 60-80 years 0.14-0.19 mg/kg, >80 years
  Arms: Bolus
Drug: Remimazolam continuous — Remimazolam 12 mg/kg/hr
  Arms: Continuous

SUMMARY:
Remimazolam is a newly introduced intravenous anesthetic, with rapid onset and offset. Although it is known to cause less hemodynamic instability, the incidence hypotension is the one of the most frequent adverse events with its use. For anesthetic induction, remimazolam can be used either as bolus dose or as continuous infusion.

This study is aimed to investigate the incidence of hypotension after anesthetic induction with bolus (0.14-0.33 mg/kg) or continuous (12 mg/kg/hr) remimazolam administration.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective surgery under general anesthesia
* adult patient (over 19 years old)
* American Society of Anesthesiology Physical Status I-III

Exclusion Criteria:

* arrythmia
* liver dysfunction
* kidney dysfunction
* uncontrolled hypertension
* uncontrolled diabetes mellitus
* allergic to benzodiazepines
* heart failure
* drug intoxication
* alcohol intoxication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 10 minutes after anesthetic induction
  Systolic pressure below 90 mmHg

SECONDARY OUTCOMES:
Incidence of bradycardia | 10 minutes after anesthetic induction
  heart rate below 40 beats per minute
The lowest systolic blood pressure | 10 minutes after anesthetic induction
  The lowest systolic blood pressure
Number of participants with vasoactive drug use | 10 minutes after anesthetic induction
  Use of vasoactive drug for the blood pressure or the heart rate management
Time to loss of consciousness | 10 minutes after anesthetic induction
  Time from drug administration to loss of consciousness
Dosage of remimazolam | 10 minutes after anesthetic induction
  Total dose or remimazolam used for anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Cho E Ah, Principal Investigator — Kangbuk Samsung Hospital

IPD SHARING:
Plan to Share IPD: Undecided